CLINICAL TRIAL: NCT06368245
Title: Durability of Supplementary Rod Constructs-SuppleMentAry Rod Technique (SMART)-for Long-segment Posterior Instrumented Spinal Fusion Procedures: A Multicenter Retrospective Comparative Study With Dual-rod Constructs
Brief Title: Durability of Suppl. Rod Constructs-SuppleMentAry Rod Technique for Long-segment Posterior Instrumented Spinal Fusions
Status: Recruiting | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: SMART
Record Dates: First submitted 2024-03-20; First posted 2024-04-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primary/revision long-segment posterior TL instrumented fusion with dual-rod constructs: The index surgery for this study is the primary or revision of long-segment posterior TL instrumented fusion using dual-rod construct.
  Interventions: Procedure: long-segment posterior TL instrumented fusion
- primary/revision long-segment posterior TL instrumented fusion with supplementary rod constructs: The index surgery for this study is the primary or revision of long-segment posterior TL instrumented fusion using either a supplementary rod construct.
  Interventions: Procedure: long-segment posterior TL instrumented fusion

INTERVENTIONS:
Procedure: long-segment posterior TL instrumented fusion — long-segment posterior TL instrumented fusion with either supplementary rod constructs or dual-rod constructs.

SUMMARY:
This is a multicenter retrospective comparative cohort study. The index surgery for this study is primary or revision long-segment posterior thoracolumbar (TL) instrumented fusion using either a supplementary rod construct or a dual-rod construct. Eligible patients who already had index surgery, will be identified for enrollment through a review of medical records of the participating surgeons at the study sites.

DETAILED DESCRIPTION:
This multicenter retrospective comparative cohort study will enroll 1244 patients, who underwent primary or revision long-segment posterior thoracolumbar (TL) instrumented fusion using either a supplementary rod construct or a dual-rod construct. By comparing two groups of patients, ie, patients treated with supplementary rod constructs vs dual-rod constructs, in the setting of long-segment posterior instrumented spinal fusion, this study aims to provide quality evidence regarding the benefits of supplementary rod constructs in reducing the risk of RFs and other mechanical complications. This study shall provide the first long-term clinical evidence on clinical outcome and benefit of supplementary rod constructs.

All participating surgeons will be asked to identify a time point, denoted as X, when they started using predominantly either supplementary rod constructs or dual-rod constructs for long-segment posterior TL instrumented spinal fusion. This time point X must be on or before December 31, 2020 (the last eligible date for the index surgery). Participating surgeons will be instructed to select the time point X to be as early within the collection window as feasible to maximize the available FU period.

Once the time point X is identified for a participating surgeon, medical records of patients treated by this surgeon will be reviewed to identify consecutive eligible patients with the index surgery done between the time point X and December 31, 2020, inclusive. In the case that an eligible patient had undergone several surgeries during this period, the first primary or revision of long-segment posterior TL instrumented fusion using either a supplementary rod construct or a dual-rod construct is defined as the index surgery.

Patients will then be grouped based on the rod constructs into either the supplementary rod construct group or dual-rod construct group.

The study has two FU periods:

* The first FU period is the first 2 years after the index surgery. The primary analysis will be done using data from the first 2 years of FU.
* The second FU period ends on December March 31, 20232024. The duration of this FU therefore ranges from 3 years and 3 months to 10 years and 3 months.

The primary study endpoint is the occurrence of the first RF within 2 years after the index surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years and older.
* Patients receiving long-segment posterior TL instrumented fusion using either supplementary rod constructs or dual-rod constructs (the index surgery).

  * Long-segment is defined as the UIV at a thoracic level and the LIV at the sacrum/ilium.
  * Supplementary rod constructs are defined as: in addition to the traditional two primary rods, at least one supplementary rod (eg, accessory rods or satellite rods) is used, and at least one supplementary rod and one primary rod (ie, at least two rods) together must span multiple (≥ 2) vertebral levels. The supplementary rod constructs do not include rods connected end-to-end or side-to-side that do not bridge multiple vertebral levels.
  * The index surgery can be a primary surgery or a revision surgery.
  * The index surgery, staged or non-staged, must use posterior spinal fusion but can be in combination with other approaches such as an anterior procedure.
* If the index surgery is a revision surgery, the primary rods must be replaced in the revision surgery, with the exception of Harrington or Luque rods which can remain in place.

  o If the Harrington or Luque rods remain in situ, they must already have the UIV at the thoracic level and the LIV at the sacrum/ilium, or an extension of the existing Harrington or Luque is performed such that the UIV is at the thoracic level and the LIV at the sacrum/ilium.
* The index surgery was performed between January 1, 2014, and December 31, 2020, inclusive.
* Minimum 3 months of FU after the index surgery.
* Ability to provide informed consent according to the IRB/EC defined and approved procedures if applicable for retrospective data analysis.

Exclusion Criteria:

* Spinal fusion performed for acute trauma (ie, ≤ 1 year of trauma).
* Spinal fusion performed for tumor.
* Spinal fusion performed for infection.
* Patients with Parkinson's Disease.
* Patients with neuromuscular disorders.
* Patients with spine malignancies requiring chemo- or radiation therapy.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent long-segment posterior thoracolumbar (TL) instrumented fusion
Sampling Method: Non-Probability Sample
Enrollment: 1244 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Rod fracture (RF) | 2 years
  Incidence of rod fracture(s)

SECONDARY OUTCOMES:
Time to rod fracture | 2 years
  Time to the first rod fracture after index surgery
Time to rod fracture | 10 years and 3 months
  Time to the first rod fracture after index surgery
Configurations of supplementary rod constructs | Baseline
  Descriptions of configurations of supplementary rod constructs
Treatment for rod fracture | 10 years and 3 months
  Descriptions of different treatment strategies for rod fractures
Recurrent RFs | 10 years and 3 months
  Incidence of recurrent rod fractures
Other mechanical failures | 10 years and 3 months
  Other mechanical failures other than rod fractures
Surgical complications | 10 years and 3 months
  Selective surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Justin S Smith, MD, PhD, Principal Investigator — Professor of Neurosurgery Chief of Spine Division, Fellowship Director University of Virginia
Locations (17):
- United States (9):
  - Stanford Spine Clinic, Redwood City, California
  - University of California, Sacramento, California
  - UCSF Spine Center, San Francisco, California
  - John Hopkis Hospital, Baltimore, Maryland
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - Washington University in St. Louis, School of Medicine, Saint Louis, Missouri 63110, St Louis, Missouri
  - Columbia University / NYP Och Spine Hospital, New York, New York
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - University of Calgary Spine, Calgary
  - University of Toronto, Toronto
- Duchess of Kent Children's Hospital, Hong Kong, China
- Kothari Medical Centre, Kolkata, India
- Japan (2):
  - Hamamatsu University School of Medicine, Hamamatsu
  - University of Tokyo, Tokyo
- Hospital Vall d´Hebron, Barcelona, Spain
- Acibadem Maslak Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided